CLINICAL TRIAL: NCT05563116
Title: Coronary Artery Calcium Score in People Living With HIV: the French HIV-CAC Cohort Study
Brief Title: French CAC-HIV Cohort Study
Acronym: CAC-HIV
Status: Completed | Type: Observational
Sponsor: Franck Boccara (Other)
Responsible Party: Sponsor-Investigator, Franck Boccara, Prinicipal Investigator, Senior Cardiologist, Professor of Cardiology, Saint Antoine University Hospital
Organization: Saint Antoine University Hospital (Other)
Other Study IDs: CAC-HIV
Record Dates: First submitted 2022-09-23; First posted 2022-10-03 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Calcification; HIV Infections
Keywords: Cardiovascular risk stratification; Primary cardiovascular prevention; Intermediate cardiovascular risk; France
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People living with HIV (PLHIV): Adults over 18 living with HIV. Participants were referred to one of our two study centers for cardiovascular assessment as part of their routine care.
  PLHIV are at intermediate cardiovascular risk, they present at least one cardiovascular risk factor without established cardiovascular disease.
  NB: all tests performed are part of routine care for cardiac prevention in France (no study specific interventions were performed.)
  Interventions: Diagnostic Test: Computed tomography coronary artery calcium (CAC) score (part of routine workup)
- HIV negative subjects: Adults over 18 without HIV infection. Participants were referred to one of our two study centers for cardiovascular assessment as part of their routine care.
  HIV- subjects are at intermediate cardiovascular risk, they present at least one cardiovascular risk factor without established cardiovascular disease.
  NB: all tests performed are part of routine care for cardiac prevention in France (no study specific interventions were performed.)
  Interventions: Diagnostic Test: Computed tomography coronary artery calcium (CAC) score (part of routine workup)

INTERVENTIONS:
Diagnostic Test: Computed tomography coronary artery calcium (CAC) score (part of routine workup) — Agatston method quantified coronary calcification. A prospectively ECG-triggered, non-contrasted CAC score used a non-enhanced low radiation cardiac CT scan provided onsite at both centers. Quantification of CAC was performed using a SOMATOM Definition Edge or SOMATOM Force (Siemens Medical Solutions) with standard mediastinal parameters (width, 350 Hounsfield units; level, 50 Hounsfield units), and according to the current guidelines for CAC scoring of non-contrast non-cardiac chest CT scans.
  Other Names: Non-invasive peripheral ultrasound (part of routine workup); Blood samples (part of routine workup)

SUMMARY:
Clinical study:

* Methods: observational transversal two-arm cohort study including adults living with HIV (PLHIV) and HIV negative subjects (HIV-) at intermediate cardiovascular risk. No study specific interventions were performed.
* Participants: consecutively recruited at two large public hospitals in Paris and Annecy, France where participants were referred for routine cardiac risk stratification.
* Recruitment: was from June 2013 until April 2016.
* Data: anonymous study data were collected during the ambulatory visit. No follow-up was conducted.

Study objectives:

* Primary: compare coronary artery calcification (CAC) score between PLHIV and HIV- in order to bridge gaps in current knowledge.
* Secondary: assess parameters linked to CAC score including predictors and their prevalence, association with carotid/femoral atherosclerosis, and cardiovascular risk scores (ASCVD and HEART score).

Study hypotheses:

* Primary: CAC scores would not be different between PLHIV and HIV-
* Secondary: prevalence of traditional CV risk factors would be lower in PLHIV but that HIV-related nontraditional CV risk factors (including lower grade chronic inflammation, immune dysregulation, and ARV exposure duration) would be associated with higher CAC scores and higher CV risk scores

Study Rational:

* PLHIV have an increased risk of atherosclerotic cardiovascular events compared to the general population. Primary prevention for PLHIV is important but challenging as traditional cardiovascular risk scores do not account for HIV-related factors.
* Computed tomography coronary artery calcium (CAC) score using the Agatston score is useful for detecting and quantifying coronary calcifications. In the general population, CAC score is predictive of future cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Present one or more cardiovascular risk factor
* Complete comprehensive cardiovascular assessment including a valid CAC score, vascular evaluation, interview for demographic, clinical and medical history and a medical workup.

Exclusion Criteria:

* Age younger than 18 years old
* History of established cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to one of our two study centers for cardiovascular assessment as part of their routine care.
Sampling Method: Non-Probability Sample
Enrollment: 689 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Computed tomography coronary artery calcium (CAC) score using the Agatston score | One test was performed between June 2013 and April 2016
  The investigators will measure the CAC score using the Agatston score.
  Agatston score scale: 0 (lowest risk) to >400 (severely increased risk)
  Agatston score interpretation:
  * lower scores mean lower risk
  * higher scores mean higher risk
  We will measure Agatston score then assign patients to one of four groups:
  CAC score = 0; CAC score 1-99, CAC score 100-399, CAC score > 400

SECONDARY OUTCOMES:
Distribution of cardiovascular risk factors | One assessment was performed between June 2013 and April 2016
  The investigators will measure the prevalence of traditional cardiovascular risk factors by medical interview, review of medical records and biochemical laboratory tests.
  - Traditional cardiovascular risk factors include: tobacco use, diabetes (fasting glucose and anti-diabetic drug use), hypertension (blood pressure measurement and antihypertensive drug use), lipid abnormalities (lipid panel and lipid-lowering drug use)
  We will measure the prevalence of non-traditional HIV-related cardiovascular risk factors by medical interview, medical records review and biochemical laboratory tests.
  - Non-traditional HIV-related cardiovascular risk factors include: HIV duration, antiretroviral regimen and duration, viral load, lymphocyte count and nadir.
Rate of carotid and femoral plaques | One assessment was performed between June 2013 and April 2016
  The investigators will use non-invasive ultrasound to measure carotid and femoral atherosclerosis.
Distribution of cardiovascular risk scores (ASCVD and HEART score): low, median and high level. | One assessment was performed between June 2013 and April 2016
  The investigators will calculate cardiovascular risk using the ASCVD model and the HEART model.

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous study data may be made available upon specific request, please contact Pr. Franck Boccara (franck.boccara@aphp.fr) for more information.